CLINICAL TRIAL: NCT00005618
Title: Phase II Study of Arsenic Trioxide, NSC 706363, in Relapsed of Refractory Chronic Myelogenous Leukemia
Brief Title: Arsenic Trioxide in Treating Patients With Relapsed or Refractory Chronic Myelogenous Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000067755; MSKCC-99076A; NCI-190
Record Dates: First submitted 2000-05-02; First posted 2004-04-02 (Estimated); Last update posted 2013-06-21 (Estimated); Status verified 2001-10

CONDITIONS: Leukemia
Keywords: relapsing chronic myelogenous leukemia; chronic phase chronic myelogenous leukemia; accelerated phase chronic myelogenous leukemia; blastic phase chronic myelogenous leukemia
MeSH Terms: conditions — Leukemia; Leukemia, Myeloid, Chronic-Phase; Leukemia, Myeloid, Accelerated Phase; Blast Crisis | interventions — Arsenic Trioxide

INTERVENTIONS:
Drug: arsenic trioxide

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of arsenic trioxide in treating patients who have relapsed or refractory chronic myelogenous leukemia.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the antileukemic efficacy of arsenic trioxide in patients with relapsed and/or refractory, chronic, accelerated, or blastic phase chronic myelogenous leukemia. II. Determine the pattern of clinical adverse experience in this patient population administered this drug.

OUTLINE: Patients are stratified according to disease stage (chronic phase vs accelerated phase or blastic phase). Patients receive arsenic trioxide IV over 1 hour on consecutive days or weekdays only for a total of 25 days followed by 3-5 weeks of rest. Treatment continues for a maximum of 6 courses in the absence of unacceptable toxicity or disease progression. Patients with responding disease are followed at least monthly.

PROJECTED ACCRUAL: A total of 10-27 patients will be accrued for the chronic phase stratum of this study within 2 years. A total of 17-37 patients will be accrued for the accelerated and blastic phases stratum of this study within 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Chronic myelogenous leukemia (CML) confirmed by: Cytogenetic testing demonstrating presence of t(9:22) OR RT-PCR demonstrating presence of BCR/ABL rearrangement Chronic phase Blast count less than 15% OR Accelerated phase defined by 1 or more of the following: Blast count greater than 15% but less than 30% Blast count and promyelocytes greater than 30% Basophils greater than 20% Thrombocytopenia less than 100,000/mm3 not related to therapy Cytogenetic clonal evolution (13) OR Blastic phase Blast count greater than 30% OR Evidence of extramedullary blasts Relapse from or failure to achieve a major cytogenetic response to at least 1 course of standard anti-CML therapy including interferon alfa or cytotoxic chemotherapy Must have failed adequate trial of interferon alfa unless intolerance to or contraindication to interferon alfa Not eligible for allogeneic stem cell transplant

PATIENT CHARACTERISTICS: Age: Not specified Performance status: Karnofsky 70-100% Life expectancy: Not specified Hematopoietic: See Disease Characteristics Hepatic: Bilirubin no greater than 1.5 times upper limit of normal (ULN) Renal: Creatinine no greater than 1.5 times ULN Other: Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception during and for 4 months after study No active serious infections that are not controlled by antibiotics

PRIOR CONCURRENT THERAPY: Biologic therapy: See Disease Characteristics At least 4 weeks since prior interferon alfa Chemotherapy: See Disease Characteristics At least 4 weeks since prior chemotherapy (1 day for hydroxyurea) No other concurrent chemotherapy Endocrine therapy: Not specified Radiotherapy: No concurrent radiotherapy Surgery: Not specified Other: No other concurrent investigational agents

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2000-02; Study Completion 2004-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David A. Scheinberg, MD, PhD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States